CLINICAL TRIAL: NCT00019916
Title: Vaccine Therapy With Tumor Specific p53 Peptides in Adult Patients With Adenocarcinoma of the Breast or Ovary
Brief Title: Vaccine Therapy Plus Interleukin-2 in Treating Women With Stage IV, Recurrent, or Progressive Breast or Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067279; NCI-99-C-0138; NCI-NMOB-9902; NCI-T99-0075; NCT00001828 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-12

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — aldesleukin; p53 synthetic long peptide vaccine

INTERVENTIONS:
Biological: aldesleukin
Biological: p53 peptide vaccine
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. It is not yet known whether combining vaccine therapy with interleukin-2 is effective in treating breast and ovarian cancer.

PURPOSE: This randomized phase I/II trial is studying the side effects of vaccine therapy and interleukin-2 and to see how well they work in treating women with stage IV, recurrent, or progressive breast or ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether endogenous cellular immunity to the p53 peptide vaccine is present in patients with stage IV, recurrent, or progressive breast or ovarian cancer and whether vaccination with these peptides and low-dose interleukin-2 can induce or boost the cellular immunity in these patients.
* Determine the type and characteristics of cellular immunity generated by this regimen in these patients.
* Determine the toxicity of this regimen in these patients.
* Correlate any immunologic response with any objective tumor response to this regimen in these patients.

OUTLINE: This is a randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

All patients undergo apheresis of autologous peripheral blood mononuclear cells, which are harvested and selected for monocytes on day -6. The monocyte fraction is cultured with sargramostim (GM-CSF) and interleukin-4 for 7 days and then pulsed with p53 peptide vaccine.

* Arm I: Patients receive p53 peptide vaccine subcutaneously (SC) on day 1.
* Arm II: Patients receive p53 peptide vaccine IV over 5 minutes on day 1. Treatment in both arms repeats every 3 weeks for a total of 4 vaccinations (4 courses). During courses 3 and 4, patients also receive low-dose interleukin-2 (IL-2) SC daily on days 3-7 and days 10-14. Patients with stable or responding disease may continue to receive vaccine and IL-2 treatment for up to 2 years.

Patients are followed at 1 month and then every 2-4 months for 2 years.

PROJECTED ACCRUAL: A maximum of 34 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the breast or ovary
* Stage IV, recurrent, or progressive disease with no chemotherapy or radiotherapy options available that would increase survival
* Tumor tissue available for determination of p53 protein expression and genetic mutation

  * p53-positive tumor by immunohistochemical analysis
* HLA-A2.1 positive
* No prior CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0 or 1

Life expectancy:

* More than 3 months

Hematopoietic:

* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT or SGPT no greater than 4 times normal
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No myocardial infarction within past 6 months
* No prior congestive heart failure
* No prior ventricular arrhythmias or other arrhythmias requiring therapy

Immunologic:

* Must have positive intradermal delayed hypersensitivity test for 1 of the following:

  * Mumps
  * Trichophyton
  * Tetanus
  * Candida
  * PPD
* No underlying immune deficiency
* No prior autoimmune disease including, but not limited to, the following:

  * Autoimmune neutropenia, thrombocytopenia, or hemolytic anemia
  * Systemic lupus erythematosus, Sjögren's syndrome, or scleroderma
  * Myasthenia gravis
  * Goodpasture's syndrome
  * Addison's disease
  * Hashimoto's thyroiditis
  * Active Graves' disease
* No active infection requiring antibiotics
* HIV negative

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy within the past 2 years except curatively treated carcinoma in situ of the cervix or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* At least 1 year since prior bone marrow transplantation

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Prior anticancer hormonal therapy allowed
* At least 4 weeks since prior systemic steroids and recovered

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* Chronic suppressive antibiotics allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Cellular immunity as measured by Elipsot assay and 51 Cr-release assay at baseline, and every 3 weeks

SECONDARY OUTCOMES:
Toxicity as measured by CTC v2.0 at baseline, and every 3 weeks
Tumor response as measured by CT scan at baseline, and every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Samir N. Khleif, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland